CLINICAL TRIAL: NCT03918057
Title: A Randomized Controlled Trial of Cognitive Behavioural Therapy for Insomnia in Pregnancy
Brief Title: Sleeping For Two: Trial for CBT for Insomnia in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB19-0465
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Insomnia; Sleep Disturbance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioural Therapy Group (Experimental): Participants receive 5 in-person weekly 1.5-hour sessions of cognitive-behavioural therapy for insomnia (CBT-I) for pregnant women, supervised by a registered, licensed clinical psychologist.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia
- Treatment as Usual Group (Active Comparator): Participants receive usual obstetric care and are placed on a wait-list until six months postpartum. All activities or efforts participants make to treat or improve their sleep on their own is recorded and coded. After the final assessment six months postpartum, participants have the option of receiving 1.5-hour sessions (for a total of 5 session) of cognitive-behavioural therapy for insomnia (CBT-I) for pregnant women, supervised by a registered, licensed clinical psychologist.
  Interventions: Other: Active Control

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Insomnia — Cognitive behavioural therapy for insomnia (CBT-I) is an evidence-based psychotherapeutic intervention that combines cognitive and behavioural principles. Specifically, this therapy provides psychoeducation about thoughts contributing to the maintenance of sleep problems, and instruction in behavioural techniques to help decrease sleep onset latency and promote effective sleep maintenance.
  Arms: Cognitive-Behavioural Therapy Group
Other: Active Control — Participants will receive regular obstetric care and will be placed on a wait-list for CBT-I treatment after their final assessment. All activities women try for improving their own sleep problems between assessments will be recorded and coded for.
  Arms: Treatment as Usual Group

SUMMARY:
Cognitive-behavioural therapy for insomnia (CBT-I) has been shown to be an effective treatment for insomnia in multiple populations, including women during pregnancy and postpartum. This randomized-controlled trial will compare the efficacy of CBT-I for pregnant women with insomnia to a treatment as usual group.

DETAILED DESCRIPTION:
Sleep disturbances are common during pregnancy and typically worsen as pregnancy progresses.Treating antenatal insomnia with pharmacotherapy effectively improves sleep quality and confers a protective benefit against the onset of postpartum depression; however, data suggests that pregnant women are reluctant to take prescribed medications due to perception of risk.

A large body of research has demonstrated that CBT-I has short-term efficacy equivalent to medication, while long-term results suggest that it outperforms medication. Despite the literature showing cognitive behavioural therapy for insomnia (CBT-I) to be effective in a variety of populations including postpartum women, and the demonstrated harmful consequences of sleep disturbances in late pregnancy, there have been few pilot studies examining the effectiveness of CBT-I in pregnancy, which was conducted by our group. Results suggested that CBT-I was effective and acceptable in reducing both objective and subjective indices of sleep quality and quantity of insomnia. These results are encouraging, and warrant larger investigations into the efficacy of CBT-I in pregnancy.

Research Question and Objectives:

The current proposal is an extension of a pilot study into a randomized design of in-person CBT-I compared to a treatment as usual (TAU) control for the treatment of insomnia experienced in pregnancy.

The primary aim of the current project is to evaluate the impact of a 5-week in-person CBT-I versus a control group in reducing symptoms of insomnia (assessed subjectively by self-report and objectively with actigraphy) experienced in pregnancy. The investigators hypothesize that participants who receive a 5-week program CBT-I (versus TAU) will report fewer insomnia symptoms and have improved objectively assessed sleep as measured post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* At or over the age of 18
* Between 12 and 28 weeks pregnant
* Are able to read, write and speak in English
* Have a diagnosis of insomnia according to the DSM-V criteria.

Exclusion Criteria:

* Experiencing symptoms of sleep disorders other than insomnia (i.e. restless legs syndrome [RLS], sleep-disordered breathing [SDB]
* Having a history of untreated, serious psychiatric illness (i.e., bipolar disorder, schizophrenia)
* Active suicidal ideation
* Currently taking prescribed medications for sleep problems
* Smoking, drinking alcohol or drug abuse during pregnancy
* Being pregnant with multiples
* Diagnosis of chronic pain.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up.
  The ISI is a 7-item questionnaire designed to identify cases of insomnia and evaluate treatment outcomes. The ISI assesses severity of sleep onset, sleep maintenance and early wakening problems, sleep dissatisfaction, and perceived distress caused by sleep problems. It was found to be a clinically useful tool in assessing changes in insomnia symptoms in insomnia treatment research.
Pittsburgh Sleep Quality Index | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up.
  The PSQI instrument is used in assessing one's sleep quality during the previous month. It consists of 19 self-rated items and 5 questions rated by the roommate or bed partner. There are seven components of the PSQI and these are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction.
Actigraphy (Actiwatch II, Phillips, USA) - Circadian rhythm amplitude, acrophase, mesor | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up
  Actigraphy monitoring provides objective sleep data. The values for circadian rhythm amplitude, acrophase, and mesor will be combined for each participant to describe their full Circadian rhythm.
Actigraphy (Actiwatch II, Phillips, USA) - Sleep efficiency | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up
  Actigraphy monitoring provides objective sleep data. A sleep efficiency value is recorded by the actigrapher and will be reported.
Actigraphy (Actiwatch II, Phillips, USA) - Sleep latency | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up
  Actigraphy monitoring provides objective sleep data. A sleep latency value is recorded by the actigrapher and will be reported.
Actigraphy (Actiwatch II, Phillips, USA) - Total sleep time | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up
  Actigraphy monitoring provides objective sleep data. A total sleep time value is recorded by the actigrapher and will be reported.
Actigraphy (Actiwatch II, Phillips, USA) - Number and frequency of awakenings | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up
  Actigraphy monitoring provides objective sleep data. The number of times participants wake up during nighttime sleep is recorded by the actigrapher and will be reported.
Sleep Logs - Latency | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up
  Sleep logs provide self-reported subjective sleep. One of the variables participants will report is the amount of time they think it takes them to fall asleep.
Sleep Logs - Total sleep time | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up
  Sleep logs provide self-reported subjective sleep. Participants will be asked to report on their estimated total sleep time.
Sleep Logs - Number and frequency of awakenings | Change between 3 time-points: baseline, 7-week follow-up, 6-months postpartum follow-up
  Sleep logs provide self-reported subjective sleep. Participants will be asked to report on the number of times they woke up during nighttime sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Lianne Tomfohr-Madsen, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Recognizing the importance of sharing results, data will be shared in accordance with the International Committee of Medical Journal Editors' guidelines, which state that authors share with others the deidentified individual patient data underlying results presented in the trial reports (including tables, figures, and appendices or supplementary material) no later than 6 months after publication. Data will be made available upon request to the primary investigator.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be made available no later than 6 months after publication, and will be available until study records are destroyed in accordance with research ethics board requirements (min 10 years post collection).

REFERENCES:
- [Background] MacKinnon AL, Madsen JW, Dhillon A, Keys E, Giesbrecht GF, Williamson T, Metcalfe A, Campbell T, Mrklas KJ, Tomfohr-Madsen L. Sleeping for two: study protocol for a randomized controlled trial of cognitive behavioral therapy for insomnia in pregnant women. Trials. 2021 Aug 12;22(1):532. doi: 10.1186/s13063-021-05498-w. PMID 34384459
- [Derived] MacKinnon AL, Silang K, Watts D, Kaur J, Freeman M, Dewsnap K, Keys E, Madsen JW, Giesbrecht GF, Williamson T, Metcalfe A, Campbell T, Mrklas KJ, Tomfohr-Madsen LM. Sleeping for Two: a randomized controlled trial of cognitive behavioral therapy for insomnia in pregnancy. J Clin Sleep Med. 2025 Feb 1;21(2):365-376. doi: 10.5664/jcsm.11396. PMID 39436396